CLINICAL TRIAL: NCT06521424
Title: The Effects of a Novel Nutritional Product on Nutrient Gaps and Gut Health in Active Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Athletic Greens International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: AG-01-0722
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Microbiome; Nutrition, Healthy; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo Controlled Design
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Maltodextrin + Flavoring
  Interventions: Dietary Supplement: Placebo
- AG1 - Nutritional Supplement (Experimental): A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Interventions: Dietary Supplement: AG1 - Nutritional Supplement

INTERVENTIONS:
Dietary Supplement: AG1 - Nutritional Supplement — A foundational nutritional supplement consisting of vitamins, minerals, probiotics, prebiotics, and whole food ingredients
  Arms: AG1 - Nutritional Supplement
Dietary Supplement: Placebo — Maltodextrin placebo
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled study of N=20 active men and women. This study to assess the effect of a novel dietary supplement on improving nutrient gaps and the gut microbiome.

ELIGIBILITY:
Inclusion Criteria:

* Provide voluntary signed and dated informed consent.
* Be in good health as determined by medical history and routine blood chemistries.
* > 1 year of resistance training experience (minimum of 2 days per week of resistance training session with free weights)
* Age between 18 and 40 yr (inclusive).
* Subject agrees to maintain existing dietary and physical activity patterns throughout the study period.
* Subject is willing and able to comply with the study protocol.

Exclusion Criteria:

* History of unstable or new-onset cardiovascular/cardiorespiratory, liver, or renal conditions.
* History of diabetes or endocrine disorder.
* History of use of medications or dietary supplements known to confound the study or its endpoints.
* Alcohol consumption (more than 2 standard alcoholic drinks per day or more than 10 drinks per week) or drug abuse or dependence within the past 6 months.
* Current smokers or smoking within the past month.
* History of hyperparathyroidism or an untreated thyroid condition.
* History of malignancy in the previous 5 years except for non-melanoma skin cancer (basal cell cancer or squamous cell cancer of the skin).
* Prior gastrointestinal bypass surgery (Lapband), etc.
* Other known gastrointestinal or metabolic conditions that might impact nutrient absorption or metabolism, e.g., short bowel syndrome, Irritable bowel syndrome (IBS), diarrheal illnesses, history of colon resection, gastro paresis, Inborn-Errors-of-Metabolism (such as PKU).
* Chronic inflammatory condition (e.g., rheumatoid arthritis, Crohn's, ulcerative colitis, Lupus, HIV/AIDS, etc.).
* Previous medical diagnosis of asthma, gout, or fibromyalgia.
* Pregnant women, women trying to become pregnant, women less than 120 days postpartum or nursing women.
* Known sensitivity to any ingredient in the test formulations as listed in the product label.
* Currently participating in another research study with an investigational product or have been in another research study in the past 30 days.
* Any other conditions that, in the opinion of the medical staff, could confound the primary endpoints or place the subject at increased risk of harm if they were to participate.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Gut Microbiome | 14 days
  Examine changes in the gut microbiome via fecal polar metabolomics measured by LC/MS
Nutrient Gaps | 14 days
  Assess nutrient gaps by dietary record assessment utilizing The Automated Self-Administered 24-hour (ASA24®) Dietary Assessment Tool

SECONDARY OUTCOMES:
Exploratory Digestive Measures | 14 days
  A Digestive Quality of Life Questionnaire (DQLQ) will be utilized to assess the effect of the interventions on participant's digestive health. Scores range from 0 to 9 with a higher score indicating worse digestion associated with quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Hofstra University, Hempstead, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided